CLINICAL TRIAL: NCT05525312
Title: Comparison of Two Strategies of One-lung Ventilation in Patients Undergoing Carcinological Lung Resection Surgery: "Open Lung" Approach With Individualized Level of Positive End-expiratory Pressure Titrated According to the Best Lung Compliance, Versus "Standard" Care: a Randomized Controlled Trial
Brief Title: Comparison of Two Strategies of One-lung Ventilation in Patients Undergoing Carcinological Lung Resection Surgery.
Acronym: I-PEEP-THO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RECHMPL19_0492
Record Dates: First submitted 2022-08-26; First posted 2022-09-01 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2023-05

CONDITIONS: Lung Diseases
Keywords: Pulmonary resection surgery; One lung ventilation; Positive end-expiratory pressure; Esophageal pressure; Transpulmonary pressure; Lung compliance; Protective ventilation; Hypoxemia; Postoperative complications
MeSH Terms: conditions — Lung Diseases; Hypoxia; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: the "standard" protective ventilation versus an "open lung" protective ventilation protocol during a pulmonary resection surgery
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Standard" protective ventilation (Other): Patients receiving a positive-end expiratory pressure (PEEP) of 5 cmH2O
  Interventions: Procedure: "Standard" protective ventilation strategy
- "Open lung" protective ventilation protocol (Experimental): Patients with a titrated positive-end expiratory pressure (PEEP) corresponding to the best lung compliance calculated with transpulmonary pressure.
  Interventions: Procedure: "Open-lung" protective ventilation strategy

INTERVENTIONS:
Procedure: "Open-lung" protective ventilation strategy — In the "open-lung" group, the positive end-tidal pressure (PEEP) is titrated to match the best lung compliance. During a "PEEP decrement trial", PEEP is decreased from 20 cmH2O to 4 cmH2O by steps of 2 cmH2O/minute, and the driving the transpulmonary pressure (PTP) is calculated at each level of PEEP. In the "open-lung" group, the targeted PEEP corresponds to the lowest driving PTP during the "PEEP decrement trial", meaning the best lung compliance. Thereafter, the PEEP is set at this level and maintained until extubation.
  Arms: "Open lung" protective ventilation protocol
Procedure: "Standard" protective ventilation strategy — In the "standard" group, the positive end-tidal pressure (PEEP) is arbitrarily set at 5 cmH2O, since this is the currently recommended level of PEEP, commonly used in control groups of previous clinical trials.
  Arms: "Standard" protective ventilation

SUMMARY:
During thoracic surgery, one-lung ventilation (OLV) is associated with hypoxemia, lung injury, and perioperative respiratory complications. The level of positive-end expiratory pressure (PEEP) to apply during OLV remains controversial. The open-lung approach consists in setting a level of PEEP corresponding to the best lung compliance, using an esophageal catheter to measure the transpulmonary pressure. This approach has been effective in laparoscopic surgeries or acute respiratory distress syndrome, but has never been evaluated in thoracic surgery.

DETAILED DESCRIPTION:
Pulmonary resection surgery plays a key role in the treatment of localized lung cancer. During thoracic surgery, lung isolation is necessary. One-lung ventilation (OLV) is associated with frequent intraoperative respiratory complications, hypoxemia or lung injury related to mechanical ventilation. Intraoperative events increase the risk of postoperative complications resulting from either hypoxemia (atrial fibrillation, delirium, acute kidney injury) or lung injury (atelectasis, pulmonary edema, pneumonia, acute respiratory distress syndrome (ARDS)).

During OLV, a protective ventilation strategy is now recommended, including a low tidal volume (VT), using the lowest fraction of inspired oxygen (FiO2) due to the toxicity of high-oxygen concentration, and recruitment maneuvers (RM). But there is no consensus on the level of positive end-tidal pressure (PEEP) to apply. A low level of PEEP increases the risk of alveolar collapse, when a too high level leads to alveolar overdistension and increases lung dead space. The PEEP is usually arbitrary fixed to 5 cmH2O for every patient, which does not take into account the individual characteristics of the patient. Recent clinical trials in thoracic surgery showed that titration of PEEP according to the lowest airway driving pressure [end-inspiratory plateau pressure - total end-expiratory pressure], compared to a standard PEEP of 5 cmH2O, increased oxygenation and lung mechanics, and decreased significantly respiratory complications.

The transpulmonary pressure (PTP) is the instantaneous difference between alveolar pressure and pleural pressure. In order to optimize the alveolocapillary gas exchange, the level of PEEP should be titrated until achieving the best lung compliance (CL), defined by the ratio [(tidal volume) / (driving PTP = end-inspiratory PTP - end-expiratory PTP)]. As the tidal volume is set on the ventilator, the level of PEEP corresponding to the best CL is the one associated with the lowest driving PTP. The "open lung" strategy consists in setting the level of PEEP according to the best CL, which is an individualized approach, probably more physiologic than the standard care.

The esophageal pressure (PES) measured by an esophageal catheter is a validated estimation of the pleural pressure. Then, the PTP could be approximated by the difference [airway plateau pressure - PES]. The placement of an esophageal catheter is safe provided that the use respects contraindications (mainly esophageal disease or varices).

In ARDS, the open lung approach using an esophageal catheter was associated with a better clinical outcome than the standard non-individualized protocol. In laparoscopic surgery, the effects of PEEP on the PTP is also well described. In thoracic surgery, to date, monitoring PES and PTP is not part of the usual care. To our knowledge, only one study described the PTP changes during OLV. In this study, the best PEEP during OLV differed from one patient to another, which goes against the "one size fits all" theory. Thus, the PEEP should be titrated and individualized. Nevertheless, the airway driving pressure is only an approximation of the PTP, since it does not take into account the pleural pressure, which is a non-negligible extra-alveolar factor when talking about patients with lung or pleural diseases. Measuring the driving PTP using an esophageal catheter is certainly more accurate.

ELIGIBILITY:
Inclusion Criteria:

* To be over 18 years old,
* To be able to attend all scheduled visits and to comply with all trial procedures,
* To be scheduled for a lung cancer resection surgery (performed by either video-assisted thoracoscopy or thoracotomy).

Exclusion Criteria:

* Non-carcinologic indication of lung resection (e.g. Lung volume reduction for bullous emphysema reduction, lung abscess),
* Bilateral pulmonary resection surgery or history of lung resection surgery,
* Lung resection under sternotomy
* Contraindication to esophageal catheter (history of esophageal varices, hepatic cirrhosis child ≥ b, esophageal or gastric surgery, thoracic radiotherapy, latex allergy),
* ASA (American Society of Anesthesiologists) score ≥ 4,
* Chronic obstructive pulmonary disease GOLD III or IV (Forced Expiratory Volume, FEV<50%),
* Uncontrolled asthma (FEV <50%),
* Intracardiac shunt,
* Hemoglobinopathy making the SpO2 values invalid,
* Heart failure NYHA III or IV,
* Documented pulmonary hypertension (Mean Pulmonary Arterial Pressure at rest, mPAP>20 mmHg),
* To be under legal protection,
* Unable to read or write,
* Lack of informed consent, or unable to give consent,
* Refusal to participate in the study,
* Pregnancy in progress or planned during the study period, pregnant or nursing women,
* Not being affiliated to a French social security system or being a beneficiary of such a system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
The incidence of intraoperative hypoxemia | During the Open-Lung Ventilation (OLV) period
  A SpO2<92% while the FiO2 is progressively decreased to 50% according to a standardized algorithm.

SECONDARY OUTCOMES:
Hypoxemia events | During the OLV period
  The number of hypoxemia events, depth, and duration of hypoxemia.
The ventilatory parameters | T1: baseline, two-lung ventilation, before OLV ; T2: 45 minutes after OLV ; T3: at the end of OLV, before re-expansion and ventilation of the operated lung ; T4: at the end of surgery, before extubation
  Plateau pressure (mbar)
The ventilatory parameters | T1: baseline, two-lung ventilation, before OLV ; T2: 45 minutes after OLV ; T3: at the end of OLV, before re-expansion and ventilation of the operated lung ; T4: at the end of surgery, before extubation
  Driving PTP (cmH2O)
The ventilatory parameters | T1: baseline, two-lung ventilation, before OLV ; T2: 45 minutes after OLV ; T3: at the end of OLV, before re-expansion and ventilation of the operated lung ; T4: at the end of surgery, before extubation
  Airway driving pressure (cmH2O)
The ventilatory parameters | T1: baseline, two-lung ventilation, before OLV ; T2: 45 minutes after OLV ; T3: at the end of OLV, before re-expansion and ventilation of the operated lung ; T4: at the end of surgery, before extubation
  Lung compliance (ml/cmH2O)
Blood gas analysis | T1: baseline, two-lung ventilation, before OLV ; T2: 45 minutes after OLV ; T3: at the end of OLV, before re-expansion and ventilation of the operated lung ; T4: at the end of surgery, before extubation
  PaO2/FiO2 ratio (mmHg)
Blood gas analysis | T1: baseline, two-lung ventilation, before OLV ; T2: 45 minutes after OLV ; T3: at the end of OLV, before re-expansion and ventilation of the operated lung ; T4: at the end of surgery, before extubation
  PaCO2 (mmHg)
Blood gas analysis | T1: baseline, two-lung ventilation, before OLV ; T2: 45 minutes after OLV ; T3: at the end of OLV, before re-expansion and ventilation of the operated lung ; T4: at the end of surgery, before extubation
  pH
Blood gas analysis | T1: baseline, two-lung ventilation, before OLV ; T2: 45 minutes after OLV ; T3: at the end of OLV, before re-expansion and ventilation of the operated lung ; T4: at the end of surgery, before extubation
  HCO3- (mmol/L)
Intraoperative events related to hypoxemia | During the OLV period
  Additional recruitment maneuvers (cmH2O)
Intraoperative events related to hypoxemia | During the OLV period
  Additional bronchoscopy
Intraoperative events related to hypoxemia | During the OLV period
  Application of a selective PEEP to the operated lung using an auxiliary valve
Intraoperative events related to hypoxemia | During the OLV period
  Re-expansion and ventilation of the operated lung performed for hypoxemia
Intraoperative events not only due to hypoxemia | During the OLV period
  Atrial fibrillation (bpm), hypotension defined by systolic arterial pressure < 90 mmHg, needs for vasopressor,
Postoperative respiratory complications until postoperative day 28 | Day 28
  Acute respiratory distress syndrome (ARDS) (diagnosed according to the Berlin definition), atelectasis or pleural effusion (documented on a postoperative chest radiograph), pneumonia (postoperative fever combined with an evocating chest radiograph, requiring antibiotics, with or without microbiologic confirmation), need for prolonged oxygen therapy (> 48 hours), need for high-flow nasal oxygen therapy, needs for postoperative invasive or noninvasive mechanical ventilation
Non-respiratory postoperative complications until postoperative day-28 (POD28) | Day 28
  Cardiovascular events such as myocardial infarction (troponin > threshold, combined with EKG modification or chest pain) or new-onset of atrial fibrillation (if the cardiac rhythm was sinus before surgery), acute kidney injury (defined by an AKIN stage ≥ 1), stroke (with CT scan or MRI confirmation) or transient ischemic attack, delirium (acutely disturbed state of mind)
The hospital stay | Day 28 and Day 90
  The in-hospital length of stay and hospital free-days at POD28, the hospital re-admission, ICU admission, and mortality at POD28 and POD90.

CONTACTS AND LOCATIONS:
Locations (1):
- Département d'Anesthésie et Réanimation Cardiothoracique - CHU Arnaud de Villeneuve, Montpellier, France